CLINICAL TRIAL: NCT00426725
Title: Protocol for Testing the Efficiency of a Device Meant to Relieve Labour Pain
Brief Title: Testing the Efficiency of a Device Meant to Relieve Labour Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ACU Medical Technologies Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ACUMT-07-KS-3811-CTIL; HTA3811
Record Dates: First submitted 2007-01-23; First posted 2007-01-25 (Estimated); Last update posted 2008-08-01 (Estimated); Status verified 2008-07

CONDITIONS: Labour Pain
Keywords: labor; pain; relief; labour; device
MeSH Terms: conditions — Labor Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): This group uses the EasyLabour device according to the protocol
  Interventions: Device: EasyLabour
- Control (No Intervention)
  Interventions: Device: EasyLabour

INTERVENTIONS:
Device: EasyLabour — According to the trial protocol

SUMMARY:
The suggested research is aimed to test the effectiveness of an external mechanical device to be applied and used by the parturient herself in pain relieving during labour . The research is to be performed in a controlled closely observed way, to ensure the safety of the involved parturient and newborn.

DETAILED DESCRIPTION:
Clinical Trial Design A prospective controlled study meant to scientifically test the feasibility of a device to alleviate labour pain.

* Every woman will sign an informed consent form.
* Guidance for proper and safe use of the device will be given by specially trained midwives.
* The study will be performed at the Laniado Hospital-Sanz Medical Center, Netanya, Israel.
* The study group will consist of 60 women, 30 in each group.
* Eligibility : Ages Eligible for study is 18 years and up.

Participants:

* The study group shall consists of 30 parturients at active labour, with contractions, demanding to receive analgesia. The device will be given, with guidance from a pre-trained midwife and under professional supervision. This study group will include also women choosing to continue using it till the application of epidural analgesia.
* The control group shall consists of 30 parturients at active labour, with contractions, choosing to receive epidural analgesia.

Inclusion criteria:

* Women with low-risk normal pregnancies.
* Healthy women, age 18 years or more.
* Single pregnancy
* At active labour, with contractions and labour pain.

Exclusion criteria:

* Women at high risk pregnancies (with Diabetes Mellitus, Arterial Hypertension, multiple fetal pregnancy, abnormal amniotic fluid index, Intra Uterine growth restriction(IUGR), or any situation which might imply placental insufficiency)
* Caesarean sections in the past
* Any contraindication to vaginal delivery (as breech presentation or Placenta Previa).
* Any active illness, abnormal body temperature, Fatigue, etc.
* Women complaining of any pain nonrelated to labour.

Criteria for taking out of the study:

Upon parturient's demand. Analgesia will be given upon parturient demand.

Method:

Parturients arriving at the delivery room and fitting the criteria will randomly divided into two groups: the study group, which will use the device, and the control group.

Intensity of pain will be measured in five different stages:

1. Before they put on the device.
2. Five minutes after starting to use the device.
3. After 30 minutes of use.
4. The device will be turned off for the duration of three consecutive contractions after which pain intensity will be measured.
5. The device will be turned on and pain intensity will be measured after 5 minutes of renewed use.

   * Pain intensity will be measured and defined by the participants using the Mosby Pain Rating Scale (see attached document).
   * The device will be attached to participants with uterine contractions with a frequency of at least 3 contractions every 10 minutes and cervical dilatation of at least 2 cm.
   * Both groups will be divided according to 3 age subgroups: 18 to 30, 31 to 40, and 41 to 45.
   * A further division will be according to BMI: below BMI 20, 20 to 25, and above a BMI of 25.

In both groups 6 indexes will be measured:

1. Comparison of pain intensity between subjects of both groups.
2. Stage of application of analgesia, epidural or other.
3. Length of second stage of birth.
4. Rate of instrumental deliveries.
5. Rate of Caesarean Sections due to non-advancement progressive labour, arrest of cervical dilatation, or arrest of fetal head descent .

Rate of fetal non reassuring monitor, like fetal deceleration or low variability.

Study length:

The study may take around one year, or till enough cases are collected in both groups.

Definition of success:

Success will be defined as proof of labour pain relief achievement, measured as a difference between the study and control groups, among participants in the study group, according to statistical criteria as are customary in similar studies. Exceptional success will be considered if statistical proof could be observed that using the device shortens delivery length of time, or, that using of the device diminishes the usage of epidural analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Women with low-risk normal pregnancies.
* Healthy women, age 18 years or more.
* Single pregnancy
* At active labour, with contractions and labour pain.

Exclusion Criteria:

* Women at high risk pregnancies (with Diabetes Mellitus, Arterial Hypertension, multiple fetal pregnancy, abnormal amniotic fluid index, Intra Uterine growth restriction(IUGR), or any situation which might imply placental insufficiency)
* Caesarean sections in the past
* Any contraindication to vaginal delivery (as breech presentation or Placenta Previa).
* Any active illness, abnormal body temperature, Fatigue, etc.
* Women complaining of any pain nonrelated to labour.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Mosby Pain Rating Scale (VAS) | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Shay Kevorkian, MD, Principal Investigator — Laniado Sanz Hospital - Netanya - Israel
Locations (1):
- Laniado Hospital - Sanz Medical Center, Netanya, Israel